CLINICAL TRIAL: NCT06683547
Title: The Impact of Ketone Monoester Intake on Post-exercise Hormonal Response During Recovery Following an Acute Bout of Resistance Exercise.
Brief Title: The Impact of Ketone Monoester Intake on Post-exercise Hormonal Responses After Resistance Exercise in Young Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Associate Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A00-M69-24B
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-01

CONDITIONS: Ketosis; Blood Hormones; Testing Effect of Intervention; Resistance Exercise; Ketone Body
Keywords: Ketone bodies; Exogenous ketone supplements; Resistance exercise; Testosterone; Anabolic hormones; Ketone monoester
MeSH Terms: conditions — Ketosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators and Outcome Accessors will be blinded to the intervention and control drinks. The drinks will be flavor matched and provided in an opaque bottle. An individual not involved with the study data collection, analysis and interpretation will be designated as a study blinder and randomizer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone Monoester (KET) (Active Comparator): Ketone monoester supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate dosed based on participants' body weight (0.36g/kg body weight).
  The nutritional beverage will be consumed twice: 30 minutes prior to the exercise workout (t = -60 min) and immediately following the completion of the exercise protocol (t = 0 min).
  Interventions: Dietary Supplement: Ketone Monoester (KET); Other: Resistance Exercise
- Placebo drink (Placebo Comparator): Flavoured water. Participants will consume this beverage twice: 30 minutes prior to the exercise workout (t = -60 min) and immediately following the completion of the exercise protocol (t = 0 min).
  Interventions: Dietary Supplement: Flavour matched placebo drink (CON); Other: Resistance Exercise

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KET) — Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight). The ketone brand name: delta G Oxford Ketone Ester.
  Arms: Ketone Monoester (KET)
Dietary Supplement: Flavour matched placebo drink (CON) — - Flavoured water (non-caloric bitter + citrus flavours)
  Arms: Placebo drink
Other: Resistance Exercise — - 5 sets of 10 repetitions of leg press and 3 sets of 12 repetitions of leg extension/leg curl 'supersets' (1 set of each back to back with no rest in between sets) at 95% of their 10-RM. Between-set rest intervals for the leg exercises will be 60 seconds.

SUMMARY:
This study investigates how orally ingested exogenous ketone monoester supplements affect circulating hormone concentrations in healthy young adult males after a single session of resistance exercise. Resistance exercise is known to stimulate an acute increase in the circulating concentration of various hormones that are involved in the regulation of muscle mass, including testosterone, growth hormone (GH), and insulin-like growth factor-1 (IGF-1).

Recently, there has been growing interest in how nutritional supplements impact these natural hormone responses at rest. One such intervention is the oral ingestion of exogenous ketone body supplements. Ketone bodies (i.e., β-hydroxybutyrate (β-HB), acetoacetate (AcAc), and acetone) are naturally occurring compounds that are normally produced by the body during prolonged fasting/starvation, or in response to a "ketogenic" diet (a diet very high in fat and very low in carbohydrates). These ketone body supplements taken in the form of a ketone monoester can quickly raise blood ketone levels without needing to change your diet.

Recent research has shown that the ingestion of exogenous ketone supplements or following a 'ketogenic diet' can alter the concentration of certain hormones measured in blood samples at rest. However, the effects of ketone monoester intake on the exercise-induced elevation in circulating hormones is yet to be explored.

Therefore, the purpose of this study is to examine how elevated β-HB, induced via the ingestion of the ketone monoester (R)-3-hydroxybutyl-(R)-3-hydroxybutyrate, affects blood concentrations of various anabolic hormones, during post-exercise recovery in healthy young adult males, compared to a placebo drink (flavoured water).

DETAILED DESCRIPTION:
A within-subject crossover design will be used for this randomized, double-blind, placebo-controlled study in healthy males to investigate the impact of ketone monoester (KET) intake on circulating (blood) concentrations of 'anabolic' and other hormones. There are two treatment arms in this crossover trial, including one KET arm and one placebo group. A total of 12 participants will be enrolled and undergo both treatment phases with a minimum 7-day washout period between lab visits.

The study will include a screening visit (Visit 1), 10-repetition maximum (10-RM) testing (visit 2), where participants' 10-RM will be determined for each exercise machine used, experimental trial (visit 3), minimum 7-day washout, followed by the phase 2 of the experimental trial (visit 4).

During the experimental trials, participants will arrive to the laboratory in an overnight fasted state, and the KET or placebo drink will then be administered following basal blood collection. Then, participants will perform a lower-body resistance exercise session consisting of 5 sets of 10 repetitions of leg press and 3 sets of 12 repetitions of leg extension/leg curl supersets at 95% of their determined 10-RM. Following exercise, another dose of the nutritional treatment will be administered.

Arterialized blood samples will then be collected at 13 postprandial timepoints during the 1-hour rested period and the 4-hour post-exercise recovery period to measure changes in plasma glucose and insulin concentration. Arterialized blood samples will also be utilized for quantitation of anabolic hormones, including testosterone, IGF-1, GH, cortisol, luteinizing hormone, sex-hormone binding globulin, dehydroepiandrosterone, estrogen, progesterone, and follicle-stimulating hormone.

Additionally, changes in capillary blood β-HB concentration will be assessed throughout the trials by collecting capillary blood samples at baseline and 11 postprandial timepoints during the 1-hour rested period and the 4-hour post-exercise recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male participants who are 18-40 years of age (inclusive).
* BMI >18.5 and <30.0 kg/m2
* Recreationally active (at least of 150 minutes of activity/week).
* Has maintained stable use of medication and supplements (which are not limited by the exclusion criteria), stable dietary and lifestyle habits, and stable body weight, for the last 3 months prior to screening and agree to maintain them throughout the study.
* Be willing to entirely avoid alcohol consumption 48 hours prior to the test days.
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

* Individuals with metabolic disorders including: Type I or Type II diabetes.
* Individuals with a history of thrombosis / cardiovascular disease, endocrine disorders
* Individuals with knee injuries (i.e., ACL injuries).
* Individuals with a positive medical history of unstable thyroid disease (i.e., hypothyroidism, hyperthyroidism, hyperparathyroidism, and hypoparathyroidism) and immune disorders.
* Individuals who have used tobacco products within the last 6 months.
* Chronic usage of medications known to modulate hormone levels (i.e. corticosteroids and hormone replacement therapy (HRT)) in the last 6 months.
* Current use of ketone supplements or adherence to a ketogenic diet.
* Formal or regular weightlifting activity within the last year.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis males
Enrollment: 12 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
Area under the curve for testosterone concentration. | Baseline and over 4 hours into the post-exercise recovery period
  Serum concentration of testosterone (nmol/l) and corresponding area under the curve (AUC), measured at baseline and over 4 hours into the post-exercise recovery period.
Time-course data for testosterone concentration. | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Serum concentration of testosterone (nmol/l) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).

SECONDARY OUTCOMES:
Area under the curve for growth hormone concentration | Baseline and over 4 hours into the post-exercise recovery period
  Serum concentration of growth hormone (μmol/L) and corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for growth hormone concentration. | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of growth hormone (μmol/L) measured at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for insulin-like growth factor-1 (IGF-1) concentration | Baseline and 4 hours into the post-exercise recovery period
  Serum concentration of IGF-1 (nmol/L) and corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for IGF-1 concentration | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of IGF-1 (nmol/L) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for cortisol concentration. | Baseline and over 4 hours into the post-exercise recovery period.
  Serum concentration of cortisol (nmol/L) and its corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for cortisol concentration. | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of cortisol (nmol/L) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for luteinizing hormone concentration | Baseline and 4 hours into the post-exercise recovery period
  Serum concentration of luteinizing hormone concentrations (IU/L) and corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for luteinizing hormone concentration | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of luteinizing hormone concentrations (IU/L) measured at13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for dehydroepiandrosterone (DHEA) concentration | Baseline and 4 hours into the post-exercise recovery period.
  Serum concentration of DHEA (μmol/L) and corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for DHEA concentration | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of DHEA (μmol/L) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for sex hormone-binding globulin (SHBG) concentration | Baseline and over 4 hours into the post-exercise recovery period.
  Serum concentration of SHBG (nmol/L) and corresponding area under the curve (AUC), measured at baseline and during the post-exercise recovery period.
Time-course data for SHBG concentration. | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of SHBG (nmol/L) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for progesterone concentration | Baseline and over 4 hours into the post-exercise recovery period.
  Serum concentration of progesterone (nmol/L) and its corresponding area under the curve (AUC), measured at baseline and during the post-exercise recovery period.
Time-course data for progesterone concentration. | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration of progesterone (nmol/L) measured at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for estrogen concentration | Baseline and over 4 hours into the post-exercise recovery period.
  Serum estrogen concentration (pmol/mL) and corresponding area under the curve (AUC), measured at baseline and during the post-exercise recovery period.
Time-course data for estrogen concentration | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration for estrogen (pmol/mL) measured at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for follicle stimulating hormone (FSH) concentration | Baseline and over 4 hours into the post-exercise recovery period.
  Serum concentration of FSH (IU/l) and corresponding area under the curve (AUC), measured at baseline and during the post-exercise recovery period.
Time-course data for FSH concentration. | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in serum concentration for FSH (IU/l) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for glucose concentration | Baseline and 4 hours into the post-exercise recovery period
  Plasma glucose concentration (mmol/L) and its corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for glucose concentration | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in plasma glucose concentration (mmol/L) measured at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for insulin concentration | Baseline and 4 hours into the post-exercise recovery period
  Plasma concentration of insulin (pmol/L) and corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for insulin concentration | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in plasma concentration of insulin (pmol/L) measured at baseline and at 13 timepoints (t = -60, -45, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 min).
Area under the curve for β-HB concentrations | Baseline and 4 hours into the post-exercise and postprandial period
  Capillary blood β-OHB concentration (mmol/L) and corresponding area under the curve (AUC), measured at baseline and over the post-exercise recovery period.
Time-course data for β-HB concentrations | Baseline, 1 hour pre-exercise and 4-hours during the post-exercise recovery period.
  Changes in capillary blood β-HB concentrations (mmol/L) measured at 12 timepoints (t = -60, -45, -30, 0, 15, 30, 60, 90, 120, 150, 180, 240 min).

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Churchward-Venne, PhD, Principal Investigator — Department of Kinesiology and Physical Education, McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided